CLINICAL TRIAL: NCT05430334
Title: Nicotine Flux, a Potentially Powerful Tool for Regulating Nicotine Delivery From Electronic Cigarettes: Significance of Nicotine Flux to the Rate of Nicotine Delivery and Subjective Effect
Brief Title: Assess the Influence of Nicotine Flux and Nicotine Form on Subjective Effects Related to Dependency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: American University Of Beirut; 1R01DA052565-01A1 (NIH)
Record Dates: First submitted 2022-06-08; First posted 2022-06-24 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-02

CONDITIONS: Nicotine Vaping; Nicotine Dependence; Nicotine Addiction
Keywords: Nicotine; Nicotine Flux; Vaping; ENDS; Aerosol; Combustible
MeSH Terms: conditions — Vaping; Tobacco Use Disorder

STUDY DESIGN:
Intervention Model Description: Each participant will attend the lab for five different visits that differ by nicotine flux and/or form in random order.
Who Masked: Participant, Investigator
Masking Description: Each participant will attend the lab for five different visits that differ by nicotine flux and/or form in random order. All sessions will be double-blind (Participant / Investigator). The analytical chemist will be providing the investigator with e-liquid in a random order in each session for each participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Combination One - 16μg/s protonated nicotine flux (Experimental): The investigators will test the subjective effects of nicotine flux (16μg/s) coupled with one ratio of nicotine form (100% protonated). Following a one-hour observation period, participants will use Subox Mini C in a 10-puff directed (30sec inter-puff interval) bout. One hour after the first bout, participants will be instructed to puff on the device for 60-min ad libitum. Subjective measures (i.e., nicotine dependence, drug effects, product liking, and craving) will be administered 5 times/session: 5 min before and 5 min after onset of the directed bout and 5 min before, halfway into and 5 min after onset of the ad libitum bout.
  Interventions: Combination Product: e-liquid 1
- Combination Two - 32μg/s protonated nicotine flux (Experimental): The investigators will test the subjective effects of nicotine flux (32μg/s) coupled with one ratio of nicotine form (100% protonated). Following a one-hour observation period, participants will use Subox Mini C in a 10-puff directed (30sec inter-puff interval) bout. One hour after the first bout, participants will be instructed to puff on the device for 60-min ad libitum. Subjective measures (i.e., nicotine dependence, drug effects, product liking, and craving) will be administered 5 times/session: 5 min before and 5 min after onset of the directed bout and 5 min before, halfway into and 5 min after onset of the ad libitum bout.
  Interventions: Combination Product: e-liquid 2
- Combination Three - 16μg/s free base nicotine flux (Experimental): The investigators will test the subjective effects of nicotine flux (16μg/s) coupled with one ratio of nicotine form (100% free base). Following a one-hour observation period, participants will use Subox Mini C in a 10-puff directed (30sec inter-puff interval) bout. One hour after the first bout, participants will be instructed to puff on the device for 60-min ad libitum. Subjective measures (i.e., nicotine dependence, drug effects, product liking, and craving) will be administered 5 times/session: 5 min before and 5 min after onset of the directed bout and 5 min before, halfway into and 5 min after onset of the ad libitum bout.
  Interventions: Combination Product: e-liquid 3
- Combination Four - 32μg/s free base nicotine flux (Experimental): The investigators will test the subjective effects of nicotine flux (32μg/s) coupled with one ratio of nicotine form (100% free base). Following a one-hour observation period, participants will use Subox Mini C in a 10-puff directed (30sec inter-puff interval) bout. One hour after the first bout, participants will be instructed to puff on the device for 60-min ad libitum. Subjective measures (i.e., nicotine dependence, drug effects, product liking, and craving) will be administered 5 times/session: 5 min before and 5 min after onset of the directed bout and 5 min before, halfway into and 5 min after onset of the ad libitum bout.
  Interventions: Combination Product: e-liquid 4
- Placebo - Combination Five - 0μg/s nicotine flux (Placebo Comparator): The investigators will test the subjective effects of nicotine flux (0μg/s) placebo. Following a one-hour observation period, participants will use Subox Mini C in a 10-puff directed (30sec inter-puff interval) bout. One hour after the first bout, participants will be instructed to puff on the device for 60-min ad libitum. Subjective measures (i.e., nicotine dependence, drug effects, product liking, and craving) will be administered 5 times/session: 5 min before and 5 min after onset of the directed bout and 5 min before, halfway into and 5 min after onset of the ad libitum bout.
  Interventions: Combination Product: e-liquid 5
- Combination six - 0 ug/s flux; high power/low power (Experimental): The investigators will test the subjective effects (perceived mouthful, perceived draw effort, and throat hit) at two power levels (20W and 40 W) with no nicotine in the liquid. Participants will alternate 10 directed puffs (30sec inter-puff interval) between two Subox Mini C devices differing only by the two power levels. Subjective measures will be administered following puff pairs 1&2, 5&6, and 9&10.
  Interventions: Combination Product: e-liquid 6
- Combination seven - 32 ug/s flux; high power/low power (Experimental): The investigators will test the subjective effects (perceived mouthful, perceived draw effort, and throat hit) at two power levels (20W and 40 W) and a constant nicotine flux of 32 ug/s. Participants will alternate 10 directed puffs (30sec inter-puff interval) between two Subox Mini C devices (20 W; 8mg/ml and 40 W;4 mg/ml). Subjective measures will be administered following puff pairs 1&2, 5&6, and 9&10.
  Interventions: Combination Product: e-liquid 7 and e-liquid 8
- Combination seven - 16 ug/s flux; high PG/VG / low PG/VG (Experimental): The investigators will test the subjective effects (perceived mouthful, perceived draw effort, and throat hit) at two PG/VG ratios (30/70 and 70/30). Participants will alternate 10 directed puffs (30sec inter-puff interval) between two Subox Mini C devices differing only by the two PG/VG ratios. Subjective measures will be administered following puff pairs 1&2, 5&6, and 9&10.
  Interventions: Combination Product: e-liquid 9 and e-liquid 10

INTERVENTIONS:
Combination Product: e-liquid 1 — 30/70 PG/VG ratio with nicotine concentration 4mg/ml protonated
  Arms: Combination One - 16μg/s protonated nicotine flux
Combination Product: e-liquid 2 — 30/70 PG/VG ratio with nicotine concentration 10mg/ml protonated
  Arms: Combination Two - 32μg/s protonated nicotine flux
Combination Product: e-liquid 3 — 30/70 PG/VG ratio with nicotine concentration 4mg/ml free base
  Arms: Combination Three - 16μg/s free base nicotine flux
Combination Product: e-liquid 4 — 30/70 PG/VG ratio with nicotine concentration 10mg/ml freebase
  Arms: Combination Four - 32μg/s free base nicotine flux
Combination Product: e-liquid 5 — 30/70 PG/VG ratio with nicotine concentration 0mg/ml (placebo)
  Arms: Placebo - Combination Five - 0μg/s nicotine flux
Combination Product: e-liquid 6 — 30/70 PG/VG ratio with nicotine concentration 0mg/ml
  Arms: Combination six - 0 ug/s flux; high power/low power
Combination Product: e-liquid 7 and e-liquid 8 — e-liquid 7: 30/70 PG/VG ratio with nicotine concentration 4mg/ml protonated e-liquid 8: 30/70 PG/VG ratio with nicotine concentration 8mg/ml protonated
  Arms: Combination seven - 32 ug/s flux; high power/low power
Combination Product: e-liquid 9 and e-liquid 10 — e-liquid 9: 30/70 PG/VG ratio with nicotine concentration 4mg/ml protonated e-liquid 10: 70/30 PG/VG ratio with nicotine concentration 4mg/ml protonated
  Arms: Combination seven - 16 ug/s flux; high PG/VG / low PG/VG

SUMMARY:
Electronic nicotine delivery systems (ENDS) heat and vaporize a nicotine-containing liquid to produce an aerosol that can deliver nicotine to the blood and the brain. ENDS use has increased rapidly in the last decade, especially among youth: over 20% of US high school students are current ENDS users, and there is evidence of nicotine dependence in this population. Federal legislation has been proposed that would restrict ENDS liquid nicotine concentration to make ENDS "significantly less addictive and appealing to youth." However, these and other efforts to curb addiction by limiting nicotine liquid concentration are unlikely to succeed because nicotine emissions from ENDS depend on multiple variables. To achieve the intended public health aims, regulations targeting addiction must focus on nicotine delivery, not nicotine concentration. While nicotine delivery cannot be regulated directly, the rate at which an ENDS emits nicotine, the "nicotine flux", can be regulated and, importantly, predicted based on a few device design and operating variables. However, to date there is no empirical evidence demonstrating the relationship between flux and delivery, nor between flux and the subjective effects that support nicotine dependence. Closing this gap is essential for providing an effective framework for regulating ENDS. At the American University of Beirut, the investigators will assess the relationship between nicotine flux, form, and subjective effects. Participants will use ENDS devices with varying nicotine fluxes and forms. Dependency measures, such as urge to smoke, craving, and abstinence, will be assessed. The outcome will indicate the degree to which nicotine flux/form influence subjective effects related to dependency, puffing intensity, and exposure to toxicants. In summary, this project will provide the empirical evidence needed for public health agencies to use nicotine flux as an encompassing and convenient construct to regulate nicotine delivery from ENDS.

DETAILED DESCRIPTION:
Assess the influence of nicotine flux and nicotine form on subjective effects. At AUB, the investigators will assess subjective effects (e.g. product liking, nicotine craving) and puffing topography for 130 participants who will undergo 5 ENDS use sessions (combinations 1-5) consisting of 2 bouts (10 puffs + 60min ad libitum) with 2 fluxes (16 and 32μg/s) x 2 forms (protonated, freebase) and a 0 nicotine condition. In addition, the investigators will use a state-of-the-art device to sample in situ a fraction of the aerosol generated during each puff to verify actual nicotine flux and form, and measure exposure to pulmonary toxicants (carbonyls). The investigators hypothesize that increasing nicotine flux and protonated nicotine will result in greater reductions of nicotine craving, and lower puffing intensity and carbonyl exposure. In addition, 10 participants that completed the five use sessions will attend the lab for one additional visit with the aim of determining the influence of puff-by-puff variation of ENDS power and liquid composition on puffing behavior and sensory effects. During this visit participants will complete three directed puffing bouts (10 puffs). In each bout, participants will alternate puffs between two identical ENDS devices differing by a single design factor (combinations 6-8).

ELIGIBILITY:
Inclusion Criteria:

* Must be healthy and above 18 years of age
* Must be willing to provide informed consent, attend the lab, and abstain from tobacco/nicotine as required (participants will be instructed to abstain from nicotine/tobacco and/or ENDS use for ≥12h)
* A dual ENDS and tobacco user who reports daily use of ENDS (≥ 3 mg/ml nicotine) or cigarettes (any frequency) AND someday use (≥ 3 days/week) of ENDS (≥ 3 mg/ml nicotine) or cigarettes (any frequency) for the past 3 months or longer

Exclusion Criteria:

* History of chronic disease or an uncontrolled psychiatric condition
* History of or active cardiovascular disease, low/high blood pressure, seizures, regular use of a prescription medication (except vitamins/birth control)
* Past month use of cocaine, opioids, benzodiazepines, or methamphetamines
* Individuals who report using marijuana >15/30 days
* Women will be excluded if they are breast-feeding or pregnant
* Participants intending to quit tobacco/nicotine use in the next 30 days and referred to cessation treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2022-07-13 (Actual); Primary Completion 2025-07-11 (Actual); Study Completion 2025-07-11 (Actual)

PRIMARY OUTCOMES:
Subjective Measures of Nicotine Abstinence Symptoms - PROMIS-10 Global Health measures | Visit 1 - Before starting the first session
  The PROMIS-10 Global Health measures five domains: physical function, fatigue, pain, emotional distress, and social health. 10 Items are rated on a five-point scale (Poor=1, Fair=2, Good=3, Very good=4, Excellent=5) with higher scores indicating higher activity.
Subjective Measures of Nicotine Abstinence Symptoms - The corresponding 4-item E-Cigarette Dependence | Visit 1 - Before starting the first session
  The corresponding 4-item E-Cigarette Dependence Scale that assesses dependence on ENDS. 4 Items are rated on a five-point scale (Never=1, Rarely=2, Sometimes=3, Often=4, Almost Always=5) with higher scores indicating higher activity.
Subjective Measures of Nicotine Abstinence Symptoms - The corresponding 4-item Combustible cigarette Dependence | Visit 1 - Before starting the first session
  The corresponding 4-item Combustible cigarette Dependence Scale that assesses nicotine dependence for daily and nondaily smokers. 4 Items are rated on a five-point scale (Never=1, Rarely=2, Sometimes=3, Often=4, Always=5) with higher scores indicating higher activity.
Nicotine Dependence questionnaires - The Fagerstrom Test of Nicotine Dependence | Visit 1 - Before starting the first session
  The Fagerstrom Test of Nicotine Dependence questionnaires that assesses nicotine dependence on ENDS. General questions not based on a scale.
Subjective Measures of Nicotine Abstinence Symptoms - Product liking magnitude scale | Up to 180 minutes
  Product liking will be assessed by the Electronic Cigarette Specific Effects questionnaire, general labeled magnitude scale (gLMS) on a subjective scale (0-100, not at all - extremely), with higher scores indicating higher effects.
Subjective Measures of Nicotine Abstinence Symptoms - Product liking hedonic scale | Up to 180 minutes
  Product liking will be assessed by the Electronic Cigarette Specific Effects questionnaire, general labeled hedonic scale (LHS) (0-100, most disliked sensation imaginable - most liked sensation imaginable), with higher scores indicating higher effects.
Subjective Measures of Nicotine Abstinence Symptoms - Drug Effect | Up to 180 minutes
  The Drug Effect Questionnaire (DEQ) will measure acute effects consisting of seven items: drug strength, high, feeling stimulated, good effects, bad effects, wanting more drugs, and drug liking and this will be assessed on a subjective scale (0-100, not at all-extremely), with higher scores indicating higher effects.
Subjective Measures of Nicotine Abstinence Symptoms - Smoking urges | Up to 180 minutes
  Smoking urges will be assessed by the smoking urges questionnaire on a subjective scale (0-100, Strongly disagree - strongly agree) with higher scores indicating higher urges.
Subjective Measures of Nicotine Abstinence Symptoms - Hughes and Hatsukami | Up to 180 minutes
  The Hughes-Hatsukami Withdrawal Questionnaire (HHWQ) will be assessed by the Hughes and Hatsukami 1986 questionnaire on a subjective scale (0-100, Not at all - extremely).

SECONDARY OUTCOMES:
Puff Duration | Will be measured during the approximately 5-minute, 10-puff use bout and 60-minute, ad lib use bout
  Measured topography Average Puff Duration (sec).
Flow rate | Will be measured during the approximately 5-minute, 10-puff use bout and 60-minute, ad lib use bout
  Measured topography Average Flow rate (LPM).
Puff Interval | Will be measured during the approximately 5-minute, 10-puff use bout and 60-minute, ad lib use bout
  Measured topography Average Inter Puff Interval (sec).
Number of Puffs | Will be measured during the approximately 60-minute, ad lib use bout
  Measured topography Total Number of Puffs (puffs).
Liquid consumed | Will be measured after the approximately 5-minute, 10-puff use bout and 60-minute, ad lib use bout
  Liquid consumption for each participant use session will be determined by pre- and post-weighing the ENDS device tank (g/session).
Carbonyl compound yield | Will be measured after the 60-minute, ad lib use bout
  Total Carbonyls Compounds will be quantified (microg/session).
Nicotine flux | Will be measured after the approximately 5-minute, 10-puff use bout and 60-minute, ad lib use bout
  Nicotine flux will be quantified (mg/sec).
Sensory Feedback - Perceived Mouthful | Will be measured during the approximately 5-minute, 10-puff use bout
  The perceived mouthful will be assessed using the following question: "How would you rate the amount of smoke filling your mouth during the puff you just smoked?". A subjective visual analog scale will be used (1-5, barely any smoke- a lot of smoke) with higher scores indicating higher mouthful.
Sensory feedback - Perceived Draw Effort | Will be measured during the approximately 5-minute, 10-puff use bout
  The perceived draw effort will be assessed using the following question: " How would you rate the effort needed to draw the puff you just smoked?". A subjective visual analog scale will be used (1-5, easy- hard) with higher scores indicating harder draw effort.

CONTACTS AND LOCATIONS:
Overall Officials: Soha Talih, PhD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No
Participants data will not be available to other researchers

REFERENCES:
- [Derived] El-Hellani A, Hanna E, Sharma M, Blohowiak R, Joseph P, Eid T, Nadim H, El-Hage R, Salman R, Karaoghlanian N, Adeniji A, Salam S, Talih F, Elbejjani M, Breland A, Eissenberg T, Shihadeh A, Baldassarri SR, Talih S. Nicotine flux as a powerful tool for regulating nicotine delivery from e-cigarettes: Protocol of two complimentary randomized crossover clinical trials. PLoS One. 2023 Sep 21;18(9):e0291786. doi: 10.1371/journal.pone.0291786. eCollection 2023. PMID 37733666